CLINICAL TRIAL: NCT02828631
Title: A Comparison of McGrath, Pentax and Macintosh Laryngoscopes for Nasotracheal Intubation in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AJIRB-MED-OBS-16-145
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Intubation Time; Intubation Difficulty Scale

ARMS (3):
- Macintosh laryngoscope (Active Comparator): Nasotracheal intubation by Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscope
- McGrath videolaryngoscope (Experimental): Nasotracheal intubation by McGrath videolaryngoscope
  Interventions: Device: McGrath videolaryngoscope
- Pentax videolaryngoscope (Experimental): Nasotracheal intubation by Pentax videolaryngoscope
  Interventions: Device: Pentax videolaryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope
  Arms: Macintosh laryngoscope
Device: McGrath videolaryngoscope
  Arms: McGrath videolaryngoscope
Device: Pentax videolaryngoscope
  Arms: Pentax videolaryngoscope

SUMMARY:
Videolaryngoscope provide better view of the larynx. This better view could improve the navigation of endotracheal tube in nasotracheal intubation. Contrast to the improved result in adult, one previous report using Glidescope in children did not show better performance than direct laryngoscope. The aim of this study is to compare the performance of McGrath, Pentax and Macintosh laryngoscope for nasotracheal intubation in children.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status class I, II

Exclusion Criteria:

* abnormality of airway
* bleeding tendency

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
time to intubation | 2 min
  Time from nasotracheal tube passing nose until confirmation of tracheal intubation by end-tidal carbon dioxide will be measured

SECONDARY OUTCOMES:
intubation difficulty scale | immediately after intubation
  Modified nasal intubation difficulty scale will be assessed : N1(intubation attempts), N2(operators to attempt intubation, N3(alternative intubation techniques or change head position), N4(glottic exposure), N5(lifting force required to expose the vocal cords), N6(optimise glottic exposure with backward, upward and right ward pressure), N7(techniques to aid intubation)

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou universitiy school of medicine, Suwon, Gyeong-gi Do, South Korea